CLINICAL TRIAL: NCT05948085
Title: A Pharmacokinetic Study of Zavegepant Intranasal in Healthy Adults Comparing Conventional Venous Blood Sampling With Patient-Centric Sampling
Brief Title: A Study to Compare Zavegepant Concentration Using Samples Collected From the Vein Versus Patient-Centric Microsampling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C5301022; NCT05948085 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Zavegepant; Migraine; Healthy Volunteers; Tasso
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zavegepant 10 mg Intranasal (IN) (Experimental): All participants will receive zavegepant 10 mg IN spray in period 1 and a butterscotch candy + zavegepant 10 mg IN spray in period 2
  Interventions: Drug: Zavegepant 10 mg IN

INTERVENTIONS:
Drug: Zavegepant 10 mg IN — All participants will receive zavegepant 10 mg IN spray in period 1 and a butterscotch candy + zavegepant 10 mg IN spray in period 2

SUMMARY:
The purpose of this clinical trial is to learn about the pharmacokinetics and safety of a drug called zavegepant from samples collected using a patient-centric device called Tasso-Plus (for liquid blood sample collection) and Tasso-M20 (for dried blood sample collection) compared to standard venous sample collection. This study consists of two periods and will enroll approximately 14 healthy participants. In period 1, half of the enrolled participants (n=7) will use Tasso-Plus, and the other 50% (n=7) will use Tasso-M20. For each participant, PK samples will be collected after zavegepant administration in period 1 using the assigned Tasso device simultaneously with collecting venous blood samples. In addition, taste assessments will be performed at time intervals of 1 (immediately after dosing), 5, 10 and 20 minutes after zavegepant IN administration. Also, if feasible, 4 Japanese participants will be enrolled among those 14 participants to evaluate the PK and safety of zavegepant IN in Japanese vs. non Japanese participants. In period 2, a butterscotch candy will be given 5 minutes before administering the zavegepant IN study intervention. Taste assessment will also be performed after zavegepant IN administration with a butterscotch candy in period 2. For taste assessment, each participant will record the sensory attributes at timed intervals of 1 (immediately after dosing), 5, 10 and 20 minutes after zavegepant administration in each period. The expected duration of participation from screening until follow-up telephone contact is approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age and older at the time of signing the informed consent document (ICD).
2. Male and female participants who are overtly healthy as determined by medical evaluation.
3. Body Mass Index (BMI) 16.0-32.0 kg/m2 and body weight ≥45.0 kg (99 lb).
4. Females must not be breastfeeding or lactating and must have a negative urine or serum pregnancy test (minimum sensitivity 25 international units per liter [IU/L] or equivalent units of human chorionic gonadotropin [HCG]) at screening. Woman/women of childbearing potential (WOCBP) must have negative urine or serum pregnancy test at admission.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Clinically significant history of nasal conditions that may affect the administration or absorption of the nasal product (eg, severe septum deviation or nasal deformity, inflammation, perforation, mucosal erosion, localized infection or ulceration, congestion, polyposis, rhinorrhea, nasal surgery within the previous 6 months, or nasal trauma).
3. Significant history of seizure disorder other than a single childhood febrile seizure (eg, epilepsy) or history of gallstone or cholecystectomy.
4. Any other medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to coronavirus disease 2019 (COVID-19) pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Use of organic anion transporting polypeptide 1B3 (OATP1B3) inhibitors within 14 days or 5 half-lives, whichever is longer, before first dosing.
6. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to investigational product (IP) dosing, administration of a biological product in the context of a clinical research study within 90 days prior to IP dosing, or concomitant participation in an investigational study involving no drug or device administration.
7. Any clinically significant abnormal laboratory test results or positive test found during medical screening. A single repeat for positive drug screen may be allowed at the discretion of the PI.
8. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination or nasal inspection beyond what is consistent with the target population.
9. Any reason that, in the opinion of the PI, would prevent the participant from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5301022

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14 participants were enrolled in this study.
Groups:
- Zavegepant: On Day 1 of Period 1, all participants received Zavegepant 10 milligrams (mg) via intranasal (IN) route (single use unidose nasal spray). Period 1 was followed by Period 2. On Day 1 of Period 2, all participants received a butterscotch candy and 5 minutes later received Zavegepant 10 mg single use unidose nasal spray. Participants were followed up 28-35 days after the second (last) dose.
Period: Treatment Period 1 (2 Days)
Arm/Group | Zavegepant
Started | 14
Completed | 14
Not Completed | 0
Period: Treatment Period 2 (2 Days)
Arm/Group | Zavegepant
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics analysis was evaluated on all enrolled participants.
Groups:
- Zavegepant: On Day 1 of Period 1, all participants received Zavegepant 10 mg via IN route (single use unidose nasal spray). Period 1 was followed by Period 2. On Day 1 of Period 2, all participants received a butterscotch candy and 5 minutes later received Zavegepant 10 mg single use unidose nasal spray. Participants were followed up 28-35 days after the second (last) dose.
Arm/Group | Zavegepant
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (14.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Zavegepant at 30 Minutes Post-dose on Day 1 of Period 1- Tasso Device Versus (vs.) Standard Venous Phlebotomy
Description: Tasso device used was Tasso-Plus (for liquid blood sample collection). In Period 1, for the treated participants pharmacokinetic (PK) samples were collected using Tasso-Plus and simultaneously standard venous phlebotomy. Data was to be reported for Tasso-Plus vs. venous phlebotomy concentrations (same participants).
Time Frame: 30 minutes post-dose on Day 1 of Period 1
Population: PK concentration analysis set: all enrolled participants who received 1 single IN dose of Zavegepant and provided at least 1 evaluable plasma concentration. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Groups:
- Tasso-Plus (Serum): Participants received Zavegepant 10 mg via IN route on Day 1 of Period 1. PK samples were collected using Tasso-Plus device.
- Venous Phlebotomy (Venous): Participants received Zavegepant 10 mg via IN route on Day 1 of Period 1. PK samples were collected using venous phlebotomy.
- Tasso-M20 (Dried Blood): Participants received Zavegepant 10 mg via IN route on Day 1 of Period 1. PK samples were collected using Tasso-M20 device.
- Standard Venous Phlebotomy (Plasma): Participants received Zavegepant 10 mg via IN route on Day 1 of Period 1. PK samples were collected using standard venous phlebotomy.
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 5 | 7
Nanograms per milliliter | 16.50 (6.0977) | 17.87 (7.3648) | 2.843 (1.8095) | 8.367 (5.0720)

2. Primary Outcome: Plasma Concentration of Zavegepant at 1 Hour Post-dose on Day 1 of Period 1- Tasso Device vs. Standard Venous Phlebotomy
Description: Tasso device used was Tasso-Plus (for liquid blood sample collection). In Period 1, for the treated participants PK samples were collected using Tasso-Plus and simultaneously standard venous phlebotomy. Data was to be reported for Tasso-Plus vs. venous phlebotomy concentrations (same participants).
Time Frame: 1-hour post-dose on Day 1 of Period 1
Population: PK concentration analysis set: all enrolled participants who received 1 single IN dose of Zavegepant and provided at least 1 evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Nanograms per milliliter | 11.56 (5.2627) | 12.73 (5.6686) | 2.278 (2.0138) | 7.083 (6.3027)

3. Primary Outcome: Plasma Concentration of Zavegepant at 2 Hours Post-dose on Day 1 of Period 1- Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: 2-hours post-dose on Day 1 of Period 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 6 | 7 | 6 | 7
Nanograms per milliliter | 6.515 (3.3114) | 6.493 (3.1807) | 1.443 (1.3173) | 3.791 (3.0525)

4. Primary Outcome: Plasma Concentration of Zavegepant at 4 Hours Post-dose on Day 1 of Period 1- Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: 4-hours post-dose on Day 1 of Period 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 6 | 7
Nanograms per milliliter | 2.603 (1.2826) | 2.830 (1.3228) | 0.8087 (0.52981) | 1.638 (1.1138)

5. Primary Outcome: Plasma Concentration of Zavegepant at 8 Hours Post-dose on Day 1 of Period 1- Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: 8-hours post-dose on Day 1 of Period 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 6 | 7
Nanograms per milliliter | 0.7659 (0.34305) | 0.8424 (0.36412) | 0.4005 (0.23037) | 0.5300 (0.33164)

6. Primary Outcome: Plasma Concentration of Zavegepant at 12 Hours Post-dose on Day 1 of Period 1- Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: 12-hours post-dose on Day 1 of Period 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Nanograms per milliliter | 0.3813 (0.16527) | 0.3969 (0.16154) | 0.3074 (0.19056) | 0.2753 (0.17468)

7. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of Zavegepant: - Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: Tasso: 0.5, 1, 2, 4, 8 and 12 hours post dose on Day 1 of Period 1; Venous: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post dose on Day 1 of Period 1
Population: PK parameter analysis set included all enrolled participants who received 1 single IN dose of Zavegepant and provided at least 1 evaluable PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Nanogram*hour per milliliter | 34.06 (57) | 37.22 (60) | NA (NA) — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were below the limit of quantification (BLQ). | NA (NA) — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.
Statistical Analysis 1: Comparison: Tasso-Plus (Serum) vs Venous Phlebotomy (Venous); Test type: Equivalence — Natural log-transformed AUCinf for Zavegepant were analyzed using a mixed effect model with blood collection method as a fixed effect and participant as a random effect; Ratio of Adjusted Means = 91.52, 90% CI 2-sided [87.07 to 96.19] — Ratio of adjusted means of test (Tasso plus) and reference (Venous Phlebotomy) and 90% CI for ratio presented in percentage

8. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of Last Quantifiable Concentration (AUClast) of Zavegepant - Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Nanogram*hour per milliliter | 32.71 (57) | 35.87 (60) | NA (NA) — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were BLQ. | NA (NA) — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.
Statistical Analysis 1: Comparison: Tasso-Plus (Serum) vs Venous Phlebotomy (Venous); Test type: Equivalence — Natural log-transformed AUClast for Zavegepant were analyzed using a mixed effect model with blood collection method as a fixed effect and participant as a random effect; Ratio of Adjusted Means = 91.19, 90% CI 2-sided [86.43 to 96.22] — [estimate comment as in outcome 7, analysis 1]

9. Primary Outcome: Maximum Plasma Concentration (Cmax) of Zavegepant - Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Nanogram per milliliter | 14.88 (64) | 16.33 (70) | NA (NA) — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were BLQ. | NA (NA) — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.
Statistical Analysis 1: Comparison: Tasso-Plus (Serum) vs Venous Phlebotomy (Venous); Test type: Equivalence — Natural log-transformed Cmax for Zavegepant were analyzed using a mixed effect model with blood collection method as a fixed effect and participant as a random effect; Ratio of Adjusted Means = 91.11, 90% CI 2-sided [86.32 to 96.18] — [estimate comment as in outcome 7, analysis 1]

10. Primary Outcome: Time for Cmax (Tmax) of Zavegepant - Tasso Device vs. Standard Venous Phlebotomy
Description: as for outcome 2
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Hours | 0.517 [0.500 to 1.03] | 0.500 [0.500 to 1.00] | NA [NA to NA] — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were BLQ. | NA [NA to NA] — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.

11. Primary Outcome: Terminal Half-Life (t1/2) of Zavegepant - Tasso Device vs. Standard Venous Phlebotomy
Description: t1/2 was calculated as loge (2) per kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Tasso device used was Tasso-Plus (for liquid blood sample collection). In Period 1, for the treated participants PK samples were collected using Tasso-Plus and simultaneously standard venous phlebotomy. Data was to be reported for Tasso-Plus vs. venous phlebotomy concentrations (same participants).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Hours | 2.914 (0.19069) | 3.819 (1.7522) | NA (NA) — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were BLQ. | NA (NA) — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.

12. Primary Outcome: Apparent Clearance (CL/F) of Zavegepant - Tasso Device vs. Standard Venous Phlebotomy
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Tasso device used was Tasso-Plus (for liquid blood sample collection). In Period 1, for the treated participants PK samples were collected using Tasso-Plus and simultaneously standard venous phlebotomy. Data was to be reported for Tasso-Plus vs. venous phlebotomy concentrations (same participants).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Liter per hour | 293.9 (57) | 268.9 (60) | NA (NA) — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were BLQ. | NA (NA) — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.

13. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Zavegepant - Tasso Device vs. Standard Venous Phlebotomy
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction absorbed. Tasso device used was Tasso-Plus (for liquid blood sample collection). In Period 1, for the treated participants PK samples were collected using Tasso-Plus and simultaneously standard venous phlebotomy. Data was to be reported for Tasso-Plus vs. venous phlebotomy concentrations (same participants).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Tasso-Plus (Serum) | Venous Phlebotomy (Venous) | Tasso-M20 (Dried Blood) | Standard Venous Phlebotomy (Plasma)
Number analyzed (Participants) | 7 | 7 | 7 | 7
Liter | 1232 (56) | 1372 (65) | NA (NA) — Data could not be calculated for Tasso-M20 (dried blood) reporting arm as the values were BLQ. | NA (NA) — Data could not be calculated for standard venous phlebotomy (plasma) reporting arm as the values were BLQ.

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were defined as events from Day 1 of dosing up to 35 days post last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From Day 1 of dosing up to 35 days post last dose of study drug (up to 37 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant
Number analyzed (Participants) | 14
Participants | 9

15. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory parameters criteria: a) Hematology: neutrophils/ leukocytes less than (<) 0.8* lower limit of normal (LLN); b) Urinalysis: urine hemoglobin was more than or equal to (>=)1 and for bacteria >20.
Time Frame: During study treatment (Day 1 of Period 1 and 2, 2 days)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant
Number analyzed (Participants) | 14
Participants | 2

ADVERSE EVENTS:
Time Frame: From Day 1 of dosing up to 35 days post last dose of study drug (up to 37 days)
Arm/Group | Zavegepant
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 9/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant (N=14)
Nausea (Gastrointestinal disorders) | 2
Oral discomfort (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Scar (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT05948085/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT05948085/SAP_001.pdf